CLINICAL TRIAL: NCT06547554
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Drug-drug Interaction, Pharmacokinetic, and Safety Study of Cefiderocol in Combination With Xeruborbactam in Healthy Adult Participants
Brief Title: A DDI Study to Investigate PK and Safety of Cefiderocol in Combination With Xeruborbactam in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Shionogi Inc. (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QPEX-400
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Bacterial Infections
Keywords: beta-lactamase inhibitor
MeSH Terms: conditions — Bacterial Infections | interventions — QPX7728; Cefiderocol; Glucose; Water

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Controlled, Crossover, Ascending Single Dose Design and Randomized, Double-Blind, Controlled, Multiple Dose Design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Single Dose Cohorts (Experimental): Administered single fixed dose of Xeruborbactam
  Administered single fixed dose of Cefiderocol
  Administered single fixed dose of a combination of Xeruborbactam and Cefiderocol.
  Interventions: Drug: Xeruborbactam; Drug: Cefiderocol; Drug: Xeruborbactam/Cefiderocol
- Multiple Dose Cohort Xeruborbactam (Experimental): Administered multiple fixed doses of Xeruborbactam
  Interventions: Drug: Xeruborbactam
- Multiple Dose Cohort Cefiderocol (Experimental): Administered multiple fixed doses of Cefiderocol
  Interventions: Drug: Cefiderocol
- Multiple Dose Cohort Cefiderocol and Xeruborbactam (Experimental): Administered multiple fixed doses of a combination of Cefiderocol and Xeruborbactam.
  Interventions: Drug: Xeruborbactam/Cefiderocol
- Multiple Dose Cohort Placebo (Placebo Comparator): Administered multiple fixed volumes of a placebo comparator
  Interventions: Drug: Dextrose 5% in water
- Single Dose Cohorts Placebo (Placebo Comparator): Administered single fixed volume of a placebo comparator
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Xeruborbactam — Experimental
  Other Names: QPX7728
  Arms: Multiple Dose Cohort Xeruborbactam; Single Dose Cohorts
Drug: Cefiderocol — Experimental
  Arms: Multiple Dose Cohort Cefiderocol; Single Dose Cohorts
Drug: Xeruborbactam/Cefiderocol — A combination of Xeruborbactam and Cefiderocol.
  Arms: Multiple Dose Cohort Cefiderocol and Xeruborbactam; Single Dose Cohorts
Drug: Dextrose 5% in water — Placebo
  Arms: Multiple Dose Cohort Placebo; Single Dose Cohorts Placebo

SUMMARY:
A phase 1, randomized, double blind, placebo controlled drug-drug interaction, pharmacokinetics and safety study of cefiderocol in combination with xeruborbactam in healthy adult participants

DETAILED DESCRIPTION:
Qpex Biopharma, Inc. is developing xeruborbactam, a new boron-based beta-lactamase inhibitor with activity against both serine and metallo-beta-lactamases in combination with a beta-lactam antibiotic.

Cefiderocol is a cephalosporin antibiotic approved in the US for the treatment of complicated urinary tract infections including pyelonephritis, and hospital-acquired bacterial pneumonia and ventilator-associated bacterial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 55 years of age (inclusive) at the time of signing the informed consent.
* Body mass index (BMI) ≥ 18.5 and 32 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive)
* Subjects must be judged to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram and laboratory profile
* Voluntary consent to participate in the study.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* A subject with active drug or alcohol abuse within 2 years prior to the initial study drug administration
* Females who are pregnant or lactating
* Documented hypersensitivity reaction or anaphylaxis to any medication. History of any severe hypersensitivity, anaphylaxis, or allergic reaction to cefiderocol or any other beta-lactam antibacterial drugs, or any other excipients used in the formulation (eg, cephalosporins, penicillins, carbapenems, or monobactams)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
The incidence and nature of treatment emergent adverse events (TEAE) | up to day 17 or up to day 21
  Summarized by cohort
Number of patients with changes from baseline in safety parameters | up to day 17 or up to day 21
  Summarized by cohort
Maximum plasma concentration (Cmax) | up to day 17 or up to day 21
  Summarized by cohort
Time to maximum plasma concentration (Tmax) | up to day 17 or up to day 21
  Summarized by cohort
Area under the plasma concentration versus time curve (AUC) | up to day 17 or up to day 21
  Summarized by cohort
Terminal elimination half-life (t1/2,z) | up to day 17 or up to day 21
  Summarized by cohort
Terminal elimination rate constant (λz) | up to day 17 or up to day 21
  Summarized by cohort
Total clearance (CL) | up to day 17 or up to day 21
  Summarized by cohort
Renal clearance (CLR) | up to day 17 or up to day 21
  Summarized by cohort
Fraction of dose excreted in urine (Feu) | up to day 17 or up to day 21
  Summarized by cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis Clinic, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No